CLINICAL TRIAL: NCT00786604
Title: Continuous Glucose Monitoring in Individuals With Spinal Cord Injury
Brief Title: Glucose Study, Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Kimberly D. Anderson, Ph.D., University of California, Irvine
Other Study IDs: 2007-5484
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Those with a cervical spinal cord injury
- 2: Those with a thoracic spinal cord injury
- 3: Healthy, control group

SUMMARY:
The purpose of this research study is to find out how blood sugar levels change during the day and night in people living with spinal cord injuries (SCI) and then to compare that with people who do not have a spinal cord injury.

As people with SCI get older they become more likely to develop health problems, just like everyone else. However, SCI increases the risk of certain problems. The amount of time post-SCI can also increase the risk of certain problems. This research project will focus on identifying the patterns of changes in blood sugar levels after SCI. Sugar in the blood is the important source of energy for the body. Too much sugar in the blood is known as hyperglycemia and not enough sugar in the blood is known as hypoglycemia. Under healthy conditions, the amount of sugar in the blood is automatically regulated so that a steady level is maintained. After SCI, however, this automatic regulation is damaged. The likelihood of experiencing too much or too little blood sugar is increased. Over time, having too much blood sugar can lead to the development of diabetes. In just the opposite situation, individuals with SCI can begin to experience more frequent episodes of too little blood sugar, which can lead to acute emergency situations.

The pattern of how blood sugar levels change during a typical 24-hour time period in persons with SCI is not known. There may be unknown factors that affect blood sugar levels. In order to find out that information, this study will involve continuously monitoring blood sugar over a 3-day period in a variety of persons with SCI. A non-invasive, wireless monitoring system will be attached to the abdomen. This system records blood sugar levels every 5 minutes. The information gathered from this observational study is vital to the understanding of how SCI alters the regulation of sugar levels in the blood and to the subsequent medical management of this population.

ELIGIBILITY:
Inclusion Criteria:

1. Must be greater than 1 year post-injury.
2. Must be 18-65 years of age.
3. Must have detectable neurologic impairment resulting from a spinal cord lesion.
4. Must not have any current pressure sores.
5. Must be cognitively competent and have no concomitant brain damage.
6. Must pass a medical examination by the study physician.
7. Must be healthy.
8. Must not have any physical ailments.
9. Must be cognitively competent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-65 years old, male or female, have a neurologic deficit as a result of spinal damage, pass a medical examination by the study physician, and must speak English. The characteristics of the control group are that subjects must be 18-65 years old, male or female, healthy without any physical ailments, pass a medical examination by the physician, and must speak English.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Anderson, Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States